CLINICAL TRIAL: NCT06302972
Title: Effects of Instrument Assisted Soft Tissue Mobilization Technique Along With Comprehensive Corrective Exercise Program in Upper Cross Syndrome.
Brief Title: Effects of IASTM Along With Comprehensive Corrective Exercise Program in Upper Cross Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/01771
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Upper Cross Syndrome
Keywords: Forward head angle; Pain; ROM; Rounded Shoulder
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Pain

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to the experimental group or control group after a baseline assessment with sealed enveloped method. Each participant took a envelope that identified their group and gave it to the researchers without seeing what was written. Participants were not notified which group was assigned to.
Who Masked: Participant
Masking Description: Participants were informed that they would receive treatment either from group 1 or group 2 without indicating which group should undergo IASTM and comprehensive corrective exercise program and which group undergo only comprehensive corrective exercise program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM and CCEP (Experimental): Instrument Assisted Soft Mobilization Technique; For pectoralis major:
  Subjects will be asked to lay supine with their thorax front side exposed. In abduction, restriction or adhesions will be located using scanning and gel will be applied. IASTM also address soft tissue restrictions and pain in levator scapulae, suboccipital muscles and sternocleidomastoid muscle.
  The CCEP will be designed in three phases, including initial, improvement, and maintenance.. The exercises in appropriate muscles in correct alignment during the movement pattern, the protocol focused on improving sustained postures.
  Exercises in initial phase protocol from 10 s hold x7 to 15 s hold x 10 from roller Exercises in improvement phase protocol from 10 repetition x 5 to 15 repetition x 6 from dumbbell , thera band, swiss ball and balance board
  Interventions: Other: IASTM and CCEP
- Comprehensive Corrective Exercise Program.Type (Active Comparator): The CCEP will be designed in three phases, including initial, improvement, and maintenance. Exercises are progressed in frequency and intensity during these phases, as long as the movements are performed in a good quality. The exercises in appropriate muscles in correct alignment during the movement pattern, the protocol focused on improving sustained postures. This goal was addressed in the improvement phase when necessary tissue adaptations occurred by increasing the load of exercises. In the maintenance phase, the participant continued to do the exercises and maintain the training adaptations for two weeks. The exercises will be the same as the improvement phase without any progression in intensity and frequency.
  Exercises in initial phase protocol from 10 s hold x7 to 15 s hold x 10 from roller Exercises in improvement phase protocol from 10 repetition x 5 to 15 repetition x 6 from dumbbell , thera band, swiss ball and balance board
  Interventions: Other: Traditional treatment

INTERVENTIONS:
Other: Traditional treatment — Hot Pack will be applied at the beginning of the session for 10 minutes. Wall corner stretching exercises, neck isometric exercises and neck stretching exercises will be performed Cold pack will be applied at the end of the session for a few minutes.
  Arms: Comprehensive Corrective Exercise Program.Type
Other: IASTM and CCEP — Instrument Assisted Soft Mobilization Technique (IASTM); For pectoralis major:
  Subjects will be asked to lay supine with their thorax front side exposed. In abduction, restriction or adhesions will be located using scanning and gel will be applied. IASTM also address soft tissue restrictions and pain in levator scapulae, suboccipital muscles and sternocleidomastoid muscle.
  The Comprehensive Corrective Exercise Program (CCEP) will be designed in three phases, including initial, improvement, and maintenance.. The exercises in appropriate muscles in correct alignment during the movement pattern, the protocol focused on improving sustained postures.
  Exercises in initial phase protocol from 10 s hold x7 to 15 s hold x 10 from roller Exercises in improvement phase protocol from 10 repetition x 5 to 15 repetition x 6 from dumbbell , thera band, swiss ball and balance board
  Arms: IASTM and CCEP

SUMMARY:
This study will see the effects of IASTM along with comprehensive corrective exercise program in upper cross syndrome through their effects on pain and cervical ranges as well as postural improvement. Our study targets both male and female population. In the reference study only male population was targeted which did not show effects of both techniques on the female population though females have high stress levels which may alter results.

DETAILED DESCRIPTION:
The upper cross syndrome involves stiffness of levator scapulae, pectoralis major and upper trapezius muscles and serratus anterior, deep neck flexors, rhomboids, middle and lower trapezius and scalene muscles weakness. Numerous bodily abnormalities such as headache, early deterioration of cervical spine and loss of cervical spine curve can be brought on by this syndrome. This syndrome can also result in thoracic spine abnormality and impaired glenohumeral joint biomechanics. Upper cross syndrome develops abnormality in head, neck and shoulder and develops in upper 1⁄4 of the trunk. The underlying causative agents of Upper cross syndrome are long surgeries, weakness, female gender, disability and poor posture. It was a randomized, controlled trial, conducted among patient with upper cross syndrome with Sample size was 44 by using G- Power software. Group A will be given IASTM with Graston's tool and comprehensive corrective exercise program and Group B will receive only comprehensive corrective exercise program. The protocol will consist of 12 sessions in total with 3 sessions a week 45 minutes / session for both groups. Assessment will be at baseline then after 2 weeks after that 2 weeks home plan for exercises and then after 4 weeks assessment will be done. Only pain will be assessed on alternative days

ELIGIBILITY:
Inclusion Criteria:

Age 18-40 years.

* Diagnosed patients with the upper crossed syndrome who have chronic neck
* pain for more than 3 months.
* Having neck pain scoring more than 3 on the Numeric Pain Scale were included
* in this study.
* Any abnormality in the position and rhythm of the scapula, as measured by the Scapular dyskinesis test, having postural changes such as excessive thoracic kyphosis (≥42°), forward head (≥44°) or round shoulder (≥49°) as measured by Flexicurve and photogrammetry.
* Both male and female population will be included

Exclusion Criteria:

The subjects with any previous surgery, any type of Infection Hypersensitive skin Diabetes Mellitus type II Having Traumatic Injury Psychological disorder Manual Therapy contraindication like osteoporosis, infection, Disc- Herniation acute Inflammation, burn scars, closed /non-complicated fractures and open wound.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion Cervical (Flexion) | 4 week
  Changes from baseline,2nd week, 4th week ROM range of motion of cervical flexion was taken
ROM Cervical (Extension) | 4 Week
  Changes from baseline,2nd week, 4th week ROM range of motion of cervical extension was taken
ROM Cervical (Left Lateral Flexion) | 4 week
  Changes from baseline,2nd week, 4th week ROM range of motion of Cervical Left Lateral Flexion was taken
ROM Cervical( Right Lateral Flexion) | 4 week
  Changes from baseline,2nd week, 4th week ROM range of motion of Cervical Right Lateral flexion was taken with the help of bubble Inclinometer
ROM Cervical ( Right Rotation) | 4 week
  Changes from baseline,2nd week, 4th week ROM range of motion of Cervical Right Rotation was taken
ROM Cervical ( Left Rotation) | 4 week
  Changes from baseline,2nd week, 4th week ROM range of motion of Cervical Left Rotation was taken.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 week
  NPRS is used for pain assessment. Pain assessment will be at baseline and in week one on alternative days and then after 2nd, 3rd and 4th weeks pain will be assessed on alternative days.
Flexicurve Ruler and Photogrammetry for posture | 4 week
  Excessive thoracic kyphosis, forward head or round shoulder as measured by Flexicurve and photogrammetry. For posture correction assessment will be at baseline and then after 2 weeks and then after 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ishtiaq, MSOMPT, Principal Investigator — Riphah International university Islamabad
Locations (1):
- Maroof international Hospital and Railway Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dehdilani M, Gol MK, Hashemzadeh K. Effects of Stretching Exercises on Upper Crossed Syndrome in Women after a Coronary Artery Bypass Graft. Crescent Journal of Medical & Biological Sciences. 2019 Jul 1;6(3).
- [Background] Mahmood T, Afzal MW, Waseem I, Arif MA, Mahmood W. Comparative Effectiveness of Routine Physical Therapy with and without Instrument Assisted Soft Tissue Mobilization for Improving Pain and Disability in Patients with Neck Pain Due to Upper Crossed Syndrome. Annals of Punjab Medical College (APMC). 2022 Mar 31;16(1):45-50.
- [Background] Page P. Cervicogenic headaches: an evidence-led approach to clinical management. Int J Sports Phys Ther. 2011 Sep;6(3):254-66. PMID 22034615
- [Background] Gull M, Akbar UU, Asim HM. FREQUENCY OF CHRONIC NECK PAIN IN UPPER CROSS SYNDROME IN FEMALE SCHOOL TEACHERS. Independent Journal of Allied Health Sciences. 2018;1(01):33-8.
- [Background] Ali S, Ahmad S, Jalal Y, Shah B. Effectiveness of Stretching Exercises Versus Muscle Energy Techniques in the Management of Upper Cross Syndrome: JRCRS. 2017; 5 (1): 12-16. Journal Riphah College of Rehabilitation Sciences. 2017 Mar 10;5(1):12-6.
- [Background] El-Hafez HM, Hamdy HA, Takla MK, Ahmed SEB, Genedy AF, Abd El-Azeim ASS. Instrument-assisted soft tissue mobilisation versus stripping massage for upper trapezius myofascial trigger points. J Taibah Univ Med Sci. 2020 Mar 6;15(2):87-93. doi: 10.1016/j.jtumed.2020.01.006. eCollection 2020 Apr. PMID 32368203
- [Background] Seidi F, Bayattork M, Minoonejad H, Andersen LL, Page P. Comprehensive corrective exercise program improves alignment, muscle activation and movement pattern of men with upper crossed syndrome: randomized controlled trial. Sci Rep. 2020 Nov 26;10(1):20688. doi: 10.1038/s41598-020-77571-4. PMID 33244045